CLINICAL TRIAL: NCT04176081
Title: A Prospective, Randomized, Open-label, Multi-centre, Phase II Trial Evaluating IDC/SChLAP1 as a Biomarker for Prediction of Response to Intensified Combined Modality Treatment
Brief Title: Study of Radiation Therapy in Combination With Darolutamide + Degarelix in Intermediate Risk Prostate Cancer
Acronym: SChLAP/IDC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Prostate Cancer Canada (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SChLAP/IDC Study
Record Dates: First submitted 2019-11-06; First posted 2019-11-25 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Intraductal carcinoma; SChLAP1; Radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — darolutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Radiation Therapy Only (Active Comparator): Participants randomized to Group 1 will receive radiation therapy only.
  Interventions: Radiation: Radiation Therapy
- Group 2: Radiation Therapy + darolutamide + degarelix (Experimental): Participants randomized to Group 2 will receive radiation therapy only + darolutamide + degarelix.
  Interventions: Drug: Darolutamide; Drug: Degarelix; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Darolutamide — Darolutamide will be administered orally as a tablet. Total daily dose is 1200 mg (2 tablets of 300 mg taken twice daily) for 6 months.
  Other Names: Nubeqa; ODM-201
  Arms: Group 2: Radiation Therapy + darolutamide + degarelix
Drug: Degarelix — Degarelix is administered by subcutaneous injection. The first dose of degarelix is 240 mg followed by monthly doses of 80 mg for a total treatment duration of 6 months.
  Other Names: Firmagon
  Arms: Group 2: Radiation Therapy + darolutamide + degarelix
Radiation: Radiation Therapy — The total radiotherapy dose for all subjects will be: 36.25 Gy in 5Fx. The study will not include elective nodal irradiation. Every fraction will have 3D image guidance (i.e. cone-beam CT).

SUMMARY:
Prostate cancer (PCa) is the most frequently diagnosed cancer in men and second leading cause of cancer-related death. Men with PCa have a wide range of possible outcomes if the cancer has not spread and is classified as Intermediate-Risk PCa (IR-PCa).

The standard treatment for IR-PCa is radiation therapy (RT) with or without hormone therapy which can result in cure in some men. In other men, the cancer can come back or spread to other areas of the body. Treatment response in men with IR-PCa is highly variable. This uncertainty has led to significant under- and over-treatment.

This study aims to find out if the addition of intensive treatment (hormonal therapy: darolutamide + degarelix) to standard treatment for PCa will work better than standard treatment alone. To do this, some participants will receive hormone therapy and others will not. All participants will receive RT.

Currently, it is difficult to identify men who may require more intensive therapy. Current methods, such as using prostate specific antigen (PSA) alone, may not give the doctor enough information about who requires more intensive treatment. The researchers conducting this study believe that a particular arrangement of cancer cells [called intraductal carcinoma (IDC)] and the presence of a genetic marker called SChLAP1 can be used to identify people who would benefit from more intensive therapy.

Hormonal therapy such as with drugs called darolutamide (new drug for PCa) and Degarelix, reduce androgens (male hormones, such as testosterone) or block their effect on the cells. PCa cells require androgens to grow and divide, so removal of androgens may be effective in preventing the return of cancer following radiation therapy.

Although darolutamide has been studied in about 1000 men with PCa and seems promising and well tolerated it is considered an experimental drug, therefore it can only be used in a research study such as this one. Degarelix has been approved by Health Canada to treat PCa.

This is a phase 2, open label, randomized, controlled study and will be conducted across sites in Canada. To qualify, men must have IR-PCa and have both SChLAP1 and IDC present or both absent. Participants will be randomized to receive RT with hormone therapy or RT only. The study treatment period is 6 months for the RT + hormone therapy group. RT will take about 1-2 weeks. All participants will be followed for 5 years with multiple visits to assess safety and treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age;
* Pathologic (histologic) proven diagnosis of prostate adenocarcinoma within 180 days prior to consent;
* PSA measurement performed within 60 days prior to consent;
* IR-PCa as per National Comprehensive Cancer Network (NCCN) criteria (PSA >10 and < 20 ng/mL and/or Gleason score 7 and/or T-category T2b-T2c clinical or ultrasound);
* UIR-PCa, at least one of the following:
* 2 or 3 NCCN IR-PCa criteria;
* Gleason score 4+3;
* >50% diagnostic cores involved by adenocarcinoma;
* Clinically negative (N0) stage, as defined by pelvic-CT or pelvic-MRI within 4 months prior to consent;
* No evidence of bone metastases (M0) assessed by a bone scan within 4 months prior to consent;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* Able and willing to provide signed informed consent as per International Conference on Harmonization - Good Clinical Practices Guidelines (ICH-GCP) and applicable regulations.

Exclusion Criteria:

* Received any form of hormonal therapy such as bilateral orchiectomy, LHRH agonist/antagonist (e.g. goserelin, leuprolide, degarelix, etc.), anti-androgens (e.g. flutamide, bicalutamide, etc.), 5α-reductase inhibitors (e.g. finasteride, dutasteride, etc.) and/or estrogens within 1 year of consent;
* Received prior cytotoxic therapy for prostate cancer (e.g. taxanes, mitoxantrone);
* Currently taking medications that might cause toxicity if combined with darolutamide (see section 4.6);
* Hemoglobin < 9.0 g/dL, independent of transfusion and/or growth factors, measured within 90 days prior to consent;
* Platelet count < 100,000 × 109/μL, independent of transfusion and/or growth factors, within 90 days prior to consent;
* Serum albumin < 3.0 g/dL within 90 days prior to consent;
* Abnormal renal function, assessed within 90 days prior to consent:
* Creatinine > 2mg/dL;
* Glomerular filtration rate (GFR) ≤ 35 mL/min, estimated by Cockcroft-Gault formula or measured directly by 24 hour urine.
* Abnormal liver function assessed within 90 days prior to consent:
* Total bilirubin > 1.5 times the upper limit of normal range;
* Aminotransferases (ALT or AST) >1.5 times the upper limit of normal range;
* Currently on anticoagulant therapy for any indication (e.g. atrial fibrillation, valve replacement, pulmonary embolism, etc.);
* Any cardiac events (e.g. unstable angina, myocardial infarction and/or congestive heart failure;
* Does not agree to use highly effective method of birth control if he is having sex with a woman of childbearing potential or does not agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 4 weeks following the last dose of study drug;
* Known hypersensitivity (or known allergic reaction) to the study treatment(s) or any of its ingredients (as listed in Investigator's brochure);
* Planned initiation of alternative therapy for prostate cancer or investigational therapy;
* Participation in another interventional clinical trial during and / or within 3 months of consent for this study;
* Subject was previously randomized in this trial;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-07-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | Recurrence Free Survival will be monitored for a duration of 5 years.
  Recurrence Free Survival (RFS), with recurrence event defined as (whichever occurs first):
  * Biochemical failure defined as per Phoenix criteria (i.e., a rise in PSA by 2 ng/mL or more above the nadir PSA, confirmed by a second PSA measurement)
  * Clinical, radiographic, or pathological evidence of local, regional, or distant recurrence/metastasis
  * Initiation of salvage hormonal therapy
  * Death from any cause.

SECONDARY OUTCOMES:
Difference in RFS rates (as defined in primary outcome measure) between IDC/SChLAP1 and treatment groups. | 5 years
  To prospectively assess the role of IDC/SChLAP1 in UIR-PCa treated with curative intent radiation to predict those who derive the greatest benefit from ST-2gen-ADT.
Incidence of early biochemical failure as defined by Pheonix criteria (i.e., within first 2 years of follow-up; surrogate of lethal disease). | 5 years
  To determine the impact of ADT hormone therapy combined with radiation therapy compared to radiation therapy alone in improving rates of early failures.
Rates of positive prostate biopsies (local failure) performed at time of recurrence as per standard of care. | 5 years
  To assess the patterns of failure after ST-2gen-ADT combined with SABR compared to SABR alone.
Testosterone levels | 5 years
  To determine the effect of ST-2gen-ADT combined with SABR compared to SABR alone on the duration of castrate testosterone levels (<50 ng/dL) after treatment completion.
Changes in prostate cancer-specific HRQoL as measured by abbreviated EPIC (urinary, bowel, sexual, and hormonal domains) questionnaire, as a function of treatment assignment | 5 years
  To determine the effect of ST-2gen-ADT combined with SABR compared to SABR alone on Health Related Quality of Life (HRQOL).
Rate of maximal biochemical control, defined as 2 consecutive undetectable PSA (<0.05 ng/mL) during follow-up. | 5 years
  To determine the effect of ST-2gen-ADT combined with SABR compared to SABR alone on PSA levels.
Rates of positive molecular imaging results (local, regional and/or distant failure) performed at time of recurrence as per standard of care. | 5 years
  To assess the patterns of failure after ST-2gen-ADT combined with SABR compared to SABR alone.
Changes in prostate cancer-specific HRQoL as measured by SF-12 questionnaire, as a function of treatment assignment | 5 years
  To determine the effect of ST-2gen-ADT combined with SABR compared to SABR alone on Health Related Quality of Life (HRQOL).

OTHER OUTCOMES:
Incidence of treatment-emergent Adverse Events | 5 years
  To determine the safety of ST-2gen-ADT combined with SABR compared to SABR alone.
Tolerability of Treatment | 5 years
  To determine the tolerability of ST-2gen-ADT combined with SABR compared to SABR alone by determining the number of subjects discontinuing investigational products due to Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, MD, Principal Investigator — UHN Princess Margaret Cancer Centre; Alejandro Berlin, MD, Principal Investigator — UHN Princess Margaret Cancer Centre
Locations (1):
- UHN Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No